CLINICAL TRIAL: NCT01453621
Title: Implementation of the Pediatric Emergency Care Applied Research Network (PECARN) Traumatic Brain Injury Prediction Rules Using Computerized Clinical Decision Support: An Interrupted Time Series Trial
Brief Title: Traumatic Brain Injury - Knowledge Translation
Acronym: TBI-KT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Peter S. Dayan, Associate Professor of Clinical Pediatrics, Emergency Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAI1828; ARRA Grant #S02MC19289-01-00 (Other Grant/Funding Number: ARRA Grant #S02MC19289-01-00)
Record Dates: First submitted 2011-09-27; First posted 2011-10-18 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Traumatic Brain Injury
Keywords: prediction rules; computerized clinical decision support; traumatic brain injury; blunt head trauma
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical decision support (post-intervention phase) (Experimental): Clinicians will receive computerized clinical decision support regarding the risk of clinically important traumatic brain injury (TBI) based on the prediction rules
  Interventions: Other: Computerized clinical decision support
- Standard care (pre-intervention phase) (No Intervention): Prior to implementation of the computerized clinical decision support, we will collect data to determine the baseline rate of CT use for children with minor blunt head trauma at very low risk of clinically-important traumatic brain injuries.

INTERVENTIONS:
Other: Computerized clinical decision support — Intervention sites will receive decision support regarding whether patient meets very low risk criteria for clinically-important traumatic brain injury based on the PECARN prediction rules.
  Arms: Clinical decision support (post-intervention phase)

SUMMARY:
Blunt head trauma (BHT) accounts for >450,000 emergency department (ED) visits for children annually in the US. Fortunately, >95% of head trauma in children is minor in nature. Although most children have minor head trauma, clinicians obtain cranial CTs in 35-50% of these children, which carries a radiation risk of malignancy. Recently, the investigators conducted a study of 44,000 children in the Pediatric Emergency Care Applied Research Network (PECARN) in which the investigators developed and validated clinical prediction rules that identify which children with minor BHT are at very low risk of having clinically-important traumatic brain injuries (TBI) and, therefore, do not require a CT scan. In this proposal, the investigators aim to assess whether implementing the PECARN TBI prediction rules (one for preverbal, one for verbal children) via computerized clinical decision support (CDS) decreases the number of (unnecessary) cranial CT scans obtained by ED physicians for children with minor BHT at very low risk of clinically-important TBIs. After a two-site pilot phase to test and refine the CDS, the investigators will conduct a seven-center prospective trial. The investigators will measure cranial CT use prior to and after the intervention implementation of CDS and clinician education. The investigators will study the use of CT by practitioners for children <18 years for 12 months pre- and post-intervention.

ELIGIBILITY:
Clinicians:

Our target study population includes clinicians with training in pediatrics (particularly pediatric emergency medicine)or general emergency medicine. As clinical practice is likely to vary among physicians with different training and in different settings, we will include two types of sites for this trial:

1. Pediatric emergency departments with >80% of children cared for by pediatric emergency medicine physicians or general pediatricians.
2. General emergency departments with >80% of children cared for by general emergency medicine physicians.

Patients:

Inclusion:

* children younger than 18 years who
* sustained minor blunt blunt head trauma defined by Glasgow Coma Scale (GCS) scores of 14 or 15 on initial ED evaluation

Exclusion:

Patients who have any of the following:

* blunt head trauma > 24 hours prior
* penetrating trauma
* brain tumors
* coagulopathy
* ventriculoperitoneal shunts
* preexisting neurological disorders complicating assessment
* neuroimaging obtained at an outside hospital before transfer to a study site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28669 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in proportion of cranial CT use in children with minor blunt head trauma at very low risk of clinically important traumatic brain injuries | Baseline and 1 year post-intervention
  The investigators will assess the rate of cranial CT use pre- and post implementation of computerized clinical decision support

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Dayan, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692
- [Derived] Ballard DW, Kuppermann N, Vinson DR, Tham E, Hoffman JM, Swietlik M, Deakyne Davies SJ, Alessandrini EA, Tzimenatos L, Bajaj L, Mark DG, Offerman SR, Chettipally UK, Paterno MD, Schaeffer MH, Richards R, Casper TC, Goldberg HS, Grundmeier RW, Dayan PS; Pediatric Emergency Care Applied Research Network (PECARN); Clinical Research on Emergency Services and Treatment (CREST) Network; Partners HealthCare. Implementation of a Clinical Decision Support System for Children With Minor Blunt Head Trauma Who Are at Nonnegligible Risk for Traumatic Brain Injuries. Ann Emerg Med. 2019 May;73(5):440-451. doi: 10.1016/j.annemergmed.2018.11.011. Epub 2018 Dec 22. PMID 30583957
- [Derived] Masterson Creber RM, Dayan PS, Kuppermann N, Ballard DW, Tzimenatos L, Alessandrini E, Mistry RD, Hoffman J, Vinson DR, Bakken S; Pediatric Emergency Care Applied Research Network (PECARN) and the Clinical Research on Emergency Services and Treatments (CREST) Network. Applying the RE-AIM Framework for the Evaluation of a Clinical Decision Support Tool for Pediatric Head Trauma: A Mixed-Methods Study. Appl Clin Inform. 2018 Jul;9(3):693-703. doi: 10.1055/s-0038-1669460. Epub 2018 Sep 5. PMID 30184559
- See also: PECARN Website — http://www.pecarn.org/